CLINICAL TRIAL: NCT06729177
Title: Strategic and Interactive Signing Instruction
Brief Title: Single Case Research Design: Teacher Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 514092; 1R21DC021024-01A1 (NIH)
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-09

CONDITIONS: Teacher Practice
Keywords: Sign Language; Deaf; Teacher Training
MeSH Terms: conditions — Sign Language

STUDY DESIGN:
Intervention Model Description: This research uses the noncurrent multiple baseline design across teacher participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single Case Research Design: Teacher 1 (Experimental): The PI worked with teachers to increase SISI implementation fidelity using a nonconcurrent multiple-baseline design across teacher participants. Four teachers who served deaf children were recruited from a school for the deaf. The SISI Fidelity Tool was used to observe teachers' business-as-usual language arts instruction and to establish three stable baseline data points for each teacher. Each SISI component was scored as 1 (fully implemented), 0.5 (partially implemented), or 0 (not implemented) and reported as the percentage of components implemented.
  After baseline observations were completed, the PI provided a two-day training on SISI implementation. Teacher 1 began implementing SISI for three weeks following the training, Teacher 2 began in Week 4, and Teachers 3 and 4 began in Weeks 7 and 10, respectively.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Single Case Research Design: Teacher 2 (Experimental): The PI worked with teachers to increase SISI implementation fidelity using a nonconcurrent multiple-baseline design across teacher participants. Four teachers who served deaf children were recruited from a school for the deaf. The SISI Fidelity Tool was used to observe teachers' business-as-usual language arts instruction and to establish three stable baseline data points for each teacher. Each SISI component was scored as 1 (fully implemented), 0.5 (partially implemented), or 0 (not implemented) and reported as the percentage of components implemented.
  After baseline observations were completed, the PI provided a two-day training on SISI implementation. Teacher 1 began implementing SISI for three weeks following the training, Teacher 2 began in Week 4, and Teachers 3 and 4 began in Weeks 7 and 10, respectively.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Single Case Research Design: Teacher 3 (Experimental): The PI worked with teachers to increase SISI implementation fidelity using a nonconcurrent multiple-baseline design across teacher participants. Four teachers who served deaf children were recruited from a school for the deaf. The SISI Fidelity Tool was used to observe teachers' business-as-usual language arts instruction and to establish three stable baseline data points for each teacher. Each SISI component was scored as 1 (fully implemented), 0.5 (partially implemented), or 0 (not implemented) and reported as the percentage of components implemented.
  After baseline observations were completed, the PI provided a two-day training on SISI implementation. Teacher 1 began implementing SISI for three weeks following the training, Teacher 2 began in Week 4, and Teachers 3 and 4 began in Weeks 7 and 10, respectively.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Single Case Research Design: Teacher 4 (Experimental): The PI worked with teachers to increase SISI implementation fidelity using a nonconcurrent multiple-baseline design across teacher participants. Four teachers who served deaf children were recruited from a school for the deaf. The SISI Fidelity Tool was used to observe teachers' business-as-usual language arts instruction and to establish three stable baseline data points for each teacher. Each SISI component was scored as 1 (fully implemented), 0.5 (partially implemented), or 0 (not implemented) and reported as the percentage of components implemented.
  After baseline observations were completed, the PI provided a two-day training on SISI implementation. Teacher 1 began implementing SISI for three weeks following the training, Teacher 2 began in Week 4, and Teachers 3 and 4 began in Weeks 7 and 10, respectively.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction

INTERVENTIONS:
Behavioral: Strategic and Interactive Signing Instruction — Evidence-based instructional methods, grounded in cognitive, sociocultural, and linguistic theories, are applied to interventions that support sign language development in deaf children.

SUMMARY:
This study examines whether a professional development program helps teachers implement Strategic and Interactive Signing Instruction (SISI) with higher fidelity. The training includes review of an intervention manual, live modeling of SISI components, and discussion of implementation expectations. Teacher fidelity is evaluated with the Strategic and Interactive Signing Instruction Fidelity Tool, which rates the extent to which core components are used during a intervention session. The study also documents how often teachers receive additional support (e.g., coaching) to understand which procedures help strengthen implementation.

DETAILED DESCRIPTION:
This project uses a nonconcurrent multiple-baseline design across four teachers who serve deaf children in a deaf education program. The goal is to examine changes in teachers' SISI implementation fidelity following training and coaching.

At baseline, the PI observes each teacher's typical language arts instruction using the SISI Fidelity Tool. Three stable data points are collected for each teacher before intervention. Every SISI component is scored as 1 (fully implemented), 0.5 (partially implemented), or 0 (not implemented), and then summarized as a percentage of components implemented.

After baseline, the PI provides a two-day training in SISI procedures. Teachers then begin implementing SISI in a staggered fashion: Teacher 1 starts immediately after training for three weeks; Teacher 2 begins in Week 4; Teachers 3 and 4 begin in Weeks 7 and 10. All instructional sessions are video-recorded and uploaded to a cloud platform, where the PI and a second rater review them for daily fidelity monitoring.

Throughout the study, the PI offers coaching as needed to support implementation. The PI also tracks children's progress on their individually targeted sign language skills to confirm that intervention adjustments are appropriate and timely. If implementation challenges arise or if data collection procedures are insufficiently clear or consistent, refinements may be made. Any refinements are put in place immediately and monitored for their influence on teacher fidelity and the feasibility of study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Teachers of the deaf working in a school for the deaf across kindergarten to 3rd grade levels

Exclusion Criteria:

* Not teachers of the deaf working in a school for the deaf across kindergarten to 3rd grade levels

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leala Holcomb, PhD, Principal Investigator — Center of Deafness
Locations (1):
- University of Tennessee, Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Under a data-sharing agreement that is in compliance with the internal policy at UTK, non-identifying data can be shared with other researchers for a minimum of 10 years on the University of Tennessee Research and Creative Exchange (TRACE). The raw data consists of videos of teachers, which will not be shared to maintain confidentiality. The processed data will be in the form of percentages for individual teachers across an academic year documented in a .csv file (Excel). Center for Open Science Foundation (OSF) is a free and open source project management tool that supports researchers throughout their entire project lifecycle. OSF also allows people to locate this data through project names, author names, and study keywords.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: December, 2026 to December, 2036
Access Criteria: Researchers may contact the principal investigator for additional supporting information not available on OSF.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four teachers from a school for the deaf were recruited.
Pre-assignment Details: All four teachers provided business-as-usual language instruction to generate baseline data before receiving training in Strategic and Interactive Signing Instruction (SISI) to implement during the intervention phase.
Groups:
- Single Case Research Design: A noncurrent multiple-baseline design across teachers was used to assess the support required for teachers to achieve proficiency in SISI implementation. The independent variable was SISI training, and the dependent variable was teacher fidelity to SISI as measured by the SISI Fidelity Tool.
Period: Overall Study
Arm/Group | Single Case Research Design
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population consisted of the four teacher participants enrolled in the single-case research design study.
Groups:
- Single Case Research Design: A noncurrent multiple baseline design across teacher participants will be utilized to assess the extent of support required by teachers to become proficient in SISI implementation. In this study, the independent variable is the SISI training, and the dependent variable is teacher fidelity to the SISI program as measured by the SISI fidelity checklist.
Arm/Group | Single Case Research Design
Number analyzed (Participants) | 4
Region of Enrollment [Number; unit: Participants] — All four teachers were recruited from a single school for the deaf in the United States.
  Participants
    United States | 4
Deaf Status [Number; unit: Participants] — The deaf status of all four participants was self-reported at baseline. Population: All participants reported deaf.
  Participants | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] — The ages of all four teacher participants was self-reported at baseline.
  Years | 38 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants] — The sex of all four participants was self-reported at baseline.
  Participants
    Female | 3
    Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race of all four participants was self-reported at baseline.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 3
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: SISI Fidelity
Description: The Strategic and Interactive Signing Instruction (SISI) Fidelity Tool is a 45-item observational checklist assessing adherence to the model-guided-independent cycle, scaffolding quality, and use of targeted ASL skills. Each item is rated from 0 to 1 (0 = not implemented, 0.5 = partially implemented, 1 = fully implemented). Scores are summed and converted to a percentage (0-100%). Higher scores indicate stronger fidelity of implementation.
Time Frame: Baseline began at the start of the school year for all participants. Because intervention start times were staggered in the multiple-baseline design, intervention duration ranged from approximately 12 to 40 weeks across participants.
Measure: Mean (Full Range); unit: Percentage of SISI practices implemented
Arm/Group | Single Case Research Design
Number analyzed (Participants) | 4
Percentage of SISI practices implemented | 80 [55 to 94]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through bi-weekly meetings with the participants during intervention phases for up to 40 weeks.
Description: Adverse events were monitored throughout the intervention period. The study involved minimal-risk professional development and intervention coaching. No adverse physical, psychological, or social events were observed.
Groups:
- Single Case Research Design: A noncurrent multiple-baseline design across teachers was used to assess the support required for teachers to achieve proficiency in SISI implementation. The independent variable was SISI training, and the dependent variable was participant fidelity to SISI as measured by the SISI Fidelity Tool.
Arm/Group | Single Case Research Design
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
This study used a multiple-baseline single-case design with four teachers. The design permits identification of functional relations between the intervention and changes in teacher behaviors; however, the small number of participants and the single-site setting restrict the extent to which results can be generalized beyond this context.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT06729177/Prot_SAP_ICF_000.pdf